CLINICAL TRIAL: NCT00272558
Title: Phase II Study of Carboplatin and Vinorelbine i.v. (Day 1) and Orally (Day 8) for Malignant Pleural Mesothelioma
Brief Title: Study of Carboplatin and Vinorelbine in Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPM phase II Carbo/VNB
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma; Chemotherapy
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Carboplatin; Vinorelbine

INTERVENTIONS:
Drug: Carboplatin and Vinorelbine

SUMMARY:
The purpose is to evaluate the activity and feasibility of a two drug regimen which is partly orally and partly intravenous in advanced pleural mesothelioma.

DETAILED DESCRIPTION:
Chemotherapy with carboplatin i.v. day one in each cycle Vinorelbine i.v. day one, and orally day 8 in each cycle, repeat new cycle every 3 weeks. Total of 6 cycles.

Endpoint is response rate, secondary endpoints survival and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified malignant pleural Mesothelioma
* Age above 18 years
* Performance status 0-2

Exclusion Criteria:

* No previous chemotherapy
* Normal renal, liver and bone marrow function

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Response

SECONDARY OUTCOMES:
Survival
Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Jens B Sorensen, MD, Study Chair — Dept. Oncology, Rigshospitalet
Locations (1):
- Dept. Oncol., Rigshospitalet, Copenhagen, Copenhagen, Denmark